CLINICAL TRIAL: NCT06564909
Title: Effect of L-Carnitine on Biomarkers of Myocardial Reperfusion Injury in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effect of L-Carnitine on Biomarkers of Myocardial Reperfusion Injury in Patients With STEMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed H. Mohamedy, Teaching assistant at clinical pharmacy department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC #268
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Reperfusion Injury, Myocardial; Myocardial Infarction
MeSH Terms: conditions — Myocardial Reperfusion Injury; Myocardial Infarction | interventions — Carnitine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): 38 STEMI patients undergoing PCI who will receive the standard of care for 4 weeks and will include the required antiplatelet (Dual Antiplatelet Therapy; DAPT), anticoagulants and anti-ischemic measures (high intensity statin, ACEI or aldosterone) as per latest guidelines recommendations.
  Interventions: Drug: The standard care for the management of myocardial infarction post PCI
- Test group (Experimental): 38 STEMI patients undergoing PCI who will receive the standard of care in addition to L-Carnitine 5 g intravenous administered as slow Iv push over 2-3 minutes (L-Carnitine 1 gm / 5 mL Injection®, MEPACO, Egypt) prior to PCI and then 2 g orally (Carnitol 500 mg®, Global Napi, Egypt) daily for 4 weeks after PCI
  Interventions: Drug: L-Carnitine; Drug: The standard care for the management of myocardial infarction post PCI

INTERVENTIONS:
Drug: L-Carnitine — L-Carnitine 5 g intravenous administered as slow IV push over 2-3 minutes (L-Carnitine 1 gm / 5 mL Injection®, MEPACO, Egypt) and Carnitol 500 mg® Oral, Global Napi, Egypt)
  Other Names: levocarnitine
  Arms: Test group
Drug: The standard care for the management of myocardial infarction post PCI — include the required antiplatelet (Dual Antiplatelet Therapy; DAPT), anticoagulants, and anti-ischemic measures (high-intensity statin, ACEI, or aldosterone) as per latest guidelines recommendations.
  Other Names: Guideline-directed medical therapy for STEMI

SUMMARY:
The study aims is to evaluate the efficacy and tolerability of L-Carnitine on biomarkers of myocardial reperfusion injury in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary PCI by the assessment of nitrotyrosine as an oxidative stress marker and Matrix metallopeptidase-2 (MMP-2) as a cardiac fibrosis marker

DETAILED DESCRIPTION:
This study aims to investigate the effects of L-Carnitine on biomarkers of myocardial reperfusion injury in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary PCI by the assessment of the following:

1. Measurement of nitrotyrosine as an oxidative stress marker and Matrix metallopeptidase-2 (MMP-2) as a cardiac fibrosis marker.
2. Assessment of The TIMI (thrombolysis in myocardial infarction) grade and Myocardial Blush Grade (MBG).
3. Echocardiography parameters

Patients and Methods:

Design: Prospective, randomized, open label, controlled clinical trial

Patients: A total of 76 STEMI patients undergoing primary PCI will be enrolled in the study and will be randomly assigned into one of 2 arms:

Group 1 (Control group) (n=38): STEMI patients undergoing PCI who will receive the standard of care Group 2 (Test group) (n= 38): STEMI patients undergoing PCI who will receive the standard of care in addition to L-Carnitine 5 g intravenous administered as slow Iv push over 2-3 minutes (L-Carnitine 1 gm / 5 mL Injection®, MEPACO, Egypt) prior to PCI and then 2 g orally (Carnitol 500 mg®, Global Napi, Egypt) daily for 4 weeks after PCI

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged >18 and < 75 years.
* STEMI patients undergoing PCI.

Exclusion Criteria:

* Patients with a recent history of myocardial infarction (MI), a previous PCI, a previous coronary artery bypass graft, or any cardiac surgery.
* A late presentation (>12 h), unsuccessful primary PCI (residual stenosis >50% in the culprit lesion after procedure),
* Pretreatment with thrombolytic or glycoprotein IIb/IIIa inhibitor therapy before primary PCI,
* Concurrent Infectious or active inflammatory disease,
* Severe liver or renal disease, (aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3x ULN or Total bilirubin > 3 x ULN), (CrCl < 60 ml/min (based on the Cockroft-Gault equation)
* Neoplasm, or hematological disorders
* Pregnant or breast-feeding patients
* Active participation in another clinical study
* Patients taking antioxidant drugs.
* History of or known allergy or intolerability to the study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the marker nitrotyrosine | 24 hours post PCI
  Measuring serum concentration of nitrotyrosine as an oxidative stress marker
Evaluation of the marker (MMP-2) | 24 hours post PCI
  Measuring serum concentration of Matrix metallopeptidase-2 (MMP-2) as a cardiac fibrosis marker.

SECONDARY OUTCOMES:
Assessment of Thrombolysis in Myocardial Infarction (TIMI) flow | 0-1 hour at the end of PCI
  Grade 0: No perfusion Grade 1: Penetration without perfusion Grade 2: Partial perfusion Grade 3: Complete perfusion
Assessment of Myocardial Blush Grade | 0-1 hour at the end of PCI
  Grade 0: No myocardial blush Grade 1: Minimal myocardial blush Grade 2: Moderate myocardial blush Grade 3: Normal myocardial blush
Incidence of ST-segment resolution >70 by ECG | 60 minutes post PCI
Echocardiography | 4 weeks
  Assessment of Left Ventricular Ejection Fraction (LVEF) and left ventricular diastolic and systolic volumes
Occurrence of Major Adverse Cardiac Events (MACE) | 4 weeks
  mortality, rehospitalization, reinfarction, arrhythmias, arrest, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt